CLINICAL TRIAL: NCT05104086
Title: Ultrasound Elastography in Differentiation of Endometriomas and Hemorrhagic Ovarian Cysts
Brief Title: Ultrasound Elastography in Diffferentiation of Endometriomas and Hemorrhagic Cysts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MS.19.09.821
Record Dates: First submitted 2021-10-08; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-09

CONDITIONS: Ovarian Endometrioma
Keywords: ultrasound elastography
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator
Masking Description: Single investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- evaluate the value of ultrasound elastography in dignosis of endometriomas (Active Comparator): evaluation of endometrioma by ultrasound elastography and will be repeated after 4 weeks
  Interventions: Device: ultrasound elastography
- evaluate the value of ultrasound elastography in ovarian hemorrhagic cysts (Active Comparator): revaluation of ovarian hemorrhagic cyst by ultrasound elastography and noticing the change of values
  Interventions: Device: ultrasound elastography

INTERVENTIONS:
Device: ultrasound elastography — strain ratio and resistivity index

SUMMARY:
To investigate the value of ultrasound elastography in differentiating endometriomas from ovarian hemorrhagic cysts

DETAILED DESCRIPTION:
The participants will be subjected to:

* Personal, Obstetric and gynecological History taking.
* Clinical examination.
* B-mode ultrasonography was performed to characterize the adnexal masses morphologically.
* Color Doppler ultrasound.
* Grayscale and elastographic ultrasound examination, which will be done using acoustic radiation force impulse (ARFI) imaging with virtual touch quantification (VTQ). Five consecutive measurements were recorded for each lesion from the region identified as the region of interest (ROI) and the median of these measurements was recorded as the shear wave velocity (SWV) value of the lesion. In virtual touch quantification (VTQ) the shear wave speed is expressed in m/s. Only numerical results will be taken into consideration.

  . Realtime elastographic and B-mode images simultaneously will appear as a two-panel image. Elastogram appeared in the region of interest (ROI) box to determine the target ovarian lesion and surrounding tissue, then elasticity colour code will be classified in 5 patterns : pattern 1, an absent or a very small hard area; pattern 2, hard area 45 per cent; pattern 4, peripheral hard and central soft areas; pattern 5, hard area occupying entire solid component with or without soft rim. Strain index will be analyzed, which will be obtained by comparing the absolute strain value of solid component of ovarian cyst with that of surrounding soft tissue.
* The invistigator will reevaluate the lesions 4 weeks after the initial assessment to see the possible changes in the size and/or configuration of the lesions with B-mode and elastographic ultrasonography.
* Lesion will be evaluated as endometriomas and referred for surgery when shows no significant changes in size and configuration.
* Hemorrhagic cyst diagnosis will be made if the lesion had resolved on follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient suspected to have endometrioma or hemorrhagic ovarian cysts.

Exclusion Criteria:

* Simple cysts which were defined as a sonolucent thin-walled (<3 mm thick) cyst larger than 3 cm in diameter without septations or papillary projections [12].
* Hemorrhagic cysts containing septations or mural nodules with detectable flow on Doppler ultrasonography

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2020-12-25 (Actual); Primary Completion 2021-11-25 (Estimated); Study Completion 2021-12-25 (Estimated)

PRIMARY OUTCOMES:
evalute the value of ultrasound elastography in differentiation in endometriomas and ovarian hemorrhagic cysts | 4 weeks
  the cut of value of strain ratio in diagnosis of endometrioma and ovarian hemorrhagic cyst

CONTACTS AND LOCATIONS:
Overall Officials: Alaa mosbah, professor, Principal Investigator — Mansoura university faculty of medicine,obestetric and gynecology department
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No